CLINICAL TRIAL: NCT01561287
Title: A Comparison of Dermal Autograft to Commercially Available Dermal Allograft in Breast Reconstruction
Brief Title: A Comparison of Dermal Autograft to AlloDerm in Breast Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: The Aesthetic Surgery Education & Research Foundation (Other)
Responsible Party: Principal Investigator, Brian Rinker, Associate Professor, Department of Surgery, University of Kentucky
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-0595-F2L
Record Dates: First submitted 2012-03-20; First posted 2012-03-23 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Mastectomy Related Lymphedema; Breast Reconstruction; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Alloderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dermal Autograft (Experimental)
  Interventions: Procedure: Dermal Autograft
- AlloDerm (Experimental)
  Interventions: Procedure: AlloDerm

INTERVENTIONS:
Procedure: Dermal Autograft — Patients in the dermal autograft group will undergo harvest of a dermal autograft from the lower abdomen at the time of mastectomy, which will be used to cover the lower pole of the tissue expander.
  Arms: Dermal Autograft
Procedure: AlloDerm — The acellular dermal matrix used in our study is AlloDerm (LifeCell Corp., Branchburg, N.J.) The AlloDerm group will consist of patients without a suitable abdomen for autografting and those who declined the dermal autograft procedure. Patients in the dermal allograft group will have placement of AlloDerm over the lower pole of the tissue expander. Patients with a lower abdominal scar and sufficient abdominal laxity for autograft harvest will be offered this technique.
  Arms: AlloDerm

SUMMARY:
Breast Cancer affects about 1 out of 8 American women. Twenty percent of breast cancer patients undergo some form of breast reconstruction. Several types of reconstructive procedures are available for appropriate patients. A reconstructive sequence consisting of a tissue expander followed by permanent implant placement is a popular choice for many women. In the past several years, acellular dermal matrices (allografts) have been used at the time of tissue expander placement to extend submuscular coverage. Reported benefits include the ability to initially fill the expander to a greater extent, improved control of the inframammary crease, and possible decrease in capsular contracture rate. Potential disadvantages of dermal allografts include foreign body reaction, incomplete tissue integration, or increased infection rates. The latter is especially worrisome, as infection in the setting of a tissue expander often necessitates the removal of the implant and interruption of the reconstructive sequence. There have been a few scattered reports of the use of dermal autografts in implant-based breast reconstruction, but they have not been widely used. Dermal autografts carry the potential benefit of improved tissue integration and lowered complication rates. However, to date there have been no studies which compare acellular dermal allograft matrices to dermal autograft for use in breast reconstruction. The objectives of this study are to compare dermal allograft to dermal autograft with respect to cost, tissue integration, patient satisfaction with scar, and complication profile in patients undergoing mastectomy followed by tissue expander/implant reconstruction.

DETAILED DESCRIPTION:
This is a retrospective comparative study of two established therapies. It is designed to enroll patients who will be undergoing breast reconstruction with tissue expanders/implants. Two groups will be created. One with patients receiving acellular dermal allograft for submuscular coverage and a second group of patients undergoing dermal autograft for submuscular coverage. Patients with a lower abdominal scar and sufficient abdominal laxity for autograft harvest will be offered this technique. The subset of these patients who elect to undergo autografting will comprise the autograft group. The allograft group will consist of the patients without a suitable abdomen for autografting and those who decline the autograft procedure. Patients in the allograft group will have placement of dermal allograft over the lower pole of the tissue expander. Patients in the autograft group will undergo harvest of a dermal autograft from the lower abdomen at the time of mastectomy, which will be used to cover the lower pole of the tissue expander. The following data will be recorded in an unidentifiable fashion: age, medical history, type of breast cancer treatment, type of reconstruction to include implant type, brand, implant size and characteristics, time of surgery including autograft harvest, and cost of overall procedure. Patients will receive routine follow-up care only, and the presence of any complications will be recorded. Per the standard reconstructive sequence for implant-based breast reconstruction, all patients will undergo a second surgical procedure under general anesthesia approximately three months following the initial surgical procedure for replacement of the tissue expander with a permanent implant and capsulotomy. At the time of this procedure, three small samples of the internal capsule will be harvested from standard locations with a 4mm biopsy punch. Histology with H/E and factor VIII staining will be performed on these samples to measure inflammation, tissue architecture, and vascular ingrowth. Comorbidities between patients with and without acellular dermal matrices will be evaluated using the Fisher exact test. Group differences for continuous variables will be assessed with the t test.

Statistical significance will be defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who underwent tissue expander/implant breast reconstruction will be included

Exclusion Criteria:

* Patients without the presence of breast cancer or with the presence of the BRCA gene will be excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Vascular Ingrowth | Three months post-surgery
  To accurately measure the neovascularization of the implants, the number of blood vessels per 40x high-power field (hpf) will be counted on the slides stained with Factor VIII. Any brown-staining endothelial cell or endothelial-cell cluster, clearly separate from adjacent microvessel and other connective-tissue elements, will be considered a single, countable microvessel. Vessel lumens, although usually present, will not be necessary for a structure to be defined as a microvessel, and red cells will not be used to define a vessel lumen.

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Rinker, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States